CLINICAL TRIAL: NCT01368016
Title: Nicotine Pharmacodynamics With a New Oral Nicotine Replacement Product and Nicotine Gum 4 mg. A Study in Healthy Smokers
Brief Title: Nicotine Pharmacodynamics With a New Oral Nicotine Replacement Therapy and Nicotine Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NICTDP2012; 2010-023268-42 (EudraCT Number)
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation; Nicotine Pharmacodynamics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental NRT (Experimental): A single 6 mg dose of an experimental Nicotine Replacement Therapy (NRT), with a 36-hour washout between visits.
  Interventions: Drug: Nicotine
- Nicotine GUM (Active Comparator): A single 4 mg dose of a marketed Nicotine Gum, with a 36-hour washout between visits.
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — A single 6 mg dose of an experimental Nicotine Replacement Therapy (NRT), with a 36-hour washout between visits
  Other Names: Not yet marketed
  Arms: Experimental NRT
Drug: Nicotine — A single 4 mg dose of a marketed Nicotine Gum, with a 36-hour washout between visits
  Other Names: Nicorette® Freshfruit gum
  Arms: Nicotine GUM

SUMMARY:
A comparison of two products for oral nicotine replacement with respect to relief of urges to smoke after single doses of nicotine.

DETAILED DESCRIPTION:
This study will be performed at two sites and two-hundred and fifty (250) healthy male and female subjects will be included. Treatments comprise single doses of an experimental Nicotine Replacement Therapy (NRT) and Nicorette Freshfruit gum 4 mg, which are chewed during 30 minutes. All subjects will be given both treatments in a crossover setting. The length of the time interval separating treatment visits, and during which no NRT must be used, will be at least 36 hours.

The subjects will abstain from smoking from 8 pm the evening before until the end of each visit. The subjects will take the gums according to instructions from the study personnel. After chewing, used gums will be collected for nicotine analysis.

Electronic diaries will be used to collect data. Urges to smoke will be scored on a 100 mm visual analogue scale (VAS) before the start of treatment and during 5 hours thereafter. Subjects will also be monitored to capture any adverse events that may occur.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, smoking more than 20 cigarettes daily during at least one year preceding inclusion.
* Body Mass Index (BMI) between 17.5 and 32.0 kg/m2 and a total body weight of at least 55.0 kg.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product within one month preceding the first dose of study medication.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 346 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC): Urges to Smoke-vs-Time | During 5 hours post-dose
  Area under urges to smoke-vs.-time curve

SECONDARY OUTCOMES:
Amount of Nicotine Released | 30 minutes
  The amount of nicotine released during product administration.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (2):
- Sweden (2):
  - Clinical Pharmacology, McNeil AB, Lund
  - Karolinska Trial Alliance (KTA), University Hospital Huddinge, Stockholm